CLINICAL TRIAL: NCT06163768
Title: Effects of Insulin Resistance in Non-diabetic Acute Coronary Syndrome Patients by the Homeostasis Model Assessment Index (HOMA2-IR)
Brief Title: Effects of Insulin Resistance in Non-diabetic Acute Coronary Syndrome Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Ngoc Minh Thu, University of Medicine and Pharmacy at Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nguyen Ngoc Minh Thu
Record Dates: First submitted 2023-11-15; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — insulin resistance factor (uremia)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- insulin (Other): This is a prospective study, without intervention in the clinical treatment plan at the hospital
  Interventions: Procedure: Insulin resistance

INTERVENTIONS:
Procedure: Insulin resistance — Steps to conduct testing and treatment according to the approved regimen at Ho Chi Minh City University of Medicine and Pharmacy Hospital. The researcher did not intervene in the treatment process.

SUMMARY:
Effects of insulin resistance in non-diabetic acute coronary syndrome patients by the homeostasis model assessment index (HOMA2-IR)

DETAILED DESCRIPTION:
Help patients know about insulin resistance. If this condition persists for a long time, it will reduce the ability to produce insulin, thereby leading to increased blood sugar levels, causing type 2 diabetes. Helping doctors have a more general view, in order to come up with a strategy more effective monitoring and treatment, preventing diabetes and cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Control group The researcher collected samples from healthy people over 18 years old who came for a health check and were concluded to have good health at the Health Examination Department of University of Medicine and Pharmacy Hospital, Ho Chi Minh City. Not falling within the exclusion criteria and agreeing to participate in the study were included in the study.
* Researchers -All patients diagnosed with Acute coronary syndrome who were over 18 years old, met the inclusion criteria and did not have exclusion criteria, and agreed to participate in the study were included in the study.

Exclusion Criteria:

* Control group

  * Patients < 18 years old.
  * History of heart disease or stroke
  * Exclude diabetic subjects
  * Exclude subjects at high risk of insulin resistance
* Researchers

  * Have diabetes or have previously been diagnosed with diabetes.
  * Patients < 18 years old.
  * The patient does not participate in follow-up examinations and does not follow up treatment at the medical facility.
  * The patient died before reaching the hospital.
  * Patients with severe medical diseases: cirrhosis, cancer, obstructive pulmonary disease chronic obstructive pulmonary disease, chronic heart failure, severe kidney failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Model HOMA-IR | January 2026
  Use SPSS software to analyze data

CONTACTS AND LOCATIONS:
Locations (1):
- Medical and Pharmaceutical University Hospital, Ho Chi Minh City, Five, Vietnam

IPD SHARING:
Plan to Share IPD: No